CLINICAL TRIAL: NCT06050681
Title: Calm Athlete: Feasibility of App-based Mindfulness Training on Collegiate Student-Athletes' Mental Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24377
Record Dates: First submitted 2023-08-24; First posted 2023-09-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Mindfulness; Mental Health Wellness
Keywords: Athlete

STUDY DESIGN:
Intervention Model Description: Single group intervention feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Intervention (Experimental): Participants will engage with a mobile application to complete 21 sessions lasting approximately 11 minutes of mindfulness training over 6 weeks.
  Interventions: Behavioral: Mindfulness Training

INTERVENTIONS:
Behavioral: Mindfulness Training — Participants will be asked to complete 21 mindfulness sessions within the Calm app on their own time and at a location of their choosing. They will be instructed to complete the '7 Days of Calm' program within the first two weeks of the intervention, the '7 Days of Managing Stress' program during weeks 3 & 4 of the intervention, and the 'Letting Go of Anxiety' program during the final two weeks of the intervention. The sessions have a mean run time of 11.76 minutes. Each 7-day program will be completed within a 2-week period, which equates to about one session every other day, but can be completed at any interval within those 2 weeks. All 21 sessions will be completed within a 6-week period.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of a mobile app-based mindfulness training program in collegiate student-athletes. The main questions it aims to answer are:

* Is a app-based mindfulness program feasible for use with collegiate student athletes?
* What, if any, benefits are seen in the mental wellbeing of collegiate student athletes following mindfulness training?

Participants will use the Calm app to complete semi-structured program of 21 mindfulness sessions over 6 weeks. Participants will complete each 8-15 minute sessions at a location and time of their choosing.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* NCAA athlete academically eligible to practice and compete in sport, and physically cleared by university sports medicine staff for participation
* Not a regular user of mindfulness meditation in the last 6 months (<4 sessions/month)
* Willingness to create an account on the Calm app and share usage data with researchers
* Fluent in English

Exclusion Criteria:

* Regular mindfulness meditation practice (>4 sessions/month)
* Not currently an NCAA eligible athlete
* Hospitalization or intensive outpatient treatment for mental illness within the past 2 years
* Not cleared by sports medicine staff to participate in sport due to injury at time of enrollment
* Not willing to download the Calm app and/or create an account
* Not willing to share app usage data with researchers
* Not fluent in English

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Feasibility- Adherence | Measured at end of 6 week intervention
  Proportion of prescribed sessions completed by enrolled participants
Feasibility- Participant Intervention Satisfaction | Measured at end of 6 week intervention
  Self rating of satisfaction of the intervention measured with a 5 point Likert scale (1=very dissatisfied, 5=very satisfied.
Feasibility- Retention | Measured at end of 6 week intervention and at 4 week follow up
  Proportion of enrolled participants that complete intervention and all assessments

SECONDARY OUTCOMES:
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Measured at baseline, at end of 6 week intervention and at 4 week follow-up
  12-item scale measuring mindfulness across 4 subscales: attention, present focus, awareness & acceptance. Min. score = 12, Max Score = 48, higher score represents greater level of mindfulness
College Student Athlete Life Stress Scale (CSALSS) | Measured at baseline, at end of 6 week intervention and at 4 week follow-up
  24-item questionnaire assessing stress specific to collegiate student-athlete's lives. 8 subscales are represented: academic requirements, sport injury, performance demand, coach relationships, training adaptation, family relationships, romantic relationships, interpersonal relationships. Min. score = 24, Max score = 144, higher score represents higher stress levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No